CLINICAL TRIAL: NCT03207503
Title: Neurobehavioral Mechanisms of Emotion Regulation in Depression Across the Adult Lifespan
Acronym: Lifespan
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00082070; R01MH113238-1 (Other Grant/Funding Number: NIMH); R01MH113238 (NIH)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDD patients: Participants ages 35-75 determined to be clinically depressed via structured clinical interview. No interventions will be administered as part of this study.
  Interventions: Procedure: fMRI
- non-MDD patients: Participants ages 35-75 determined to be lifetime free of psychiatric conditions as assessed by structured clinical interview. No interventions will be administered as part of this study.
  Interventions: Procedure: fMRI

INTERVENTIONS:
Procedure: fMRI — Patients will undergo fMRI imaging to assess areas of the brain that are active during emotion regulation. No clinical benefit of MRI imaging is anticipated.

SUMMARY:
The aim of this study is to test a model of demographic (age, sex), clinical, cognitive, and neurocircuitry predictors of emotion regulation ability and long-term depressive symptoms.

DETAILED DESCRIPTION:
Emotion regulation capacities are crucial for sustaining mental health in the face of cumulative stressors over one's lifetime. Although it is well documented that some emotion regulation abilities are preserved or even improved in healthy aging, little is known about why regulatory deficits persist in older adults who suffer from depression. Treatments for major depressive disorder (MDD) focus on remediating affective dysregulation processes that confer risks for disability, poor quality of life, and morbidity into late life. Theoretical perspectives on emotional aging propose myriad lifespan changes that potentially impact regulatory capacities, including structural and functional integrity of dorsal attentional and ventral affective processing pathways, cognitive status, and use of specific regulatory strategies, among others. However, there is a dearth of empirical evidence to indicate which combination of these factors critically interacts with depressive symptoms to impact emotional dysregulation in older adults, when these factors become important across the course of the adult lifespan, which strategies they apply to, and whether they can predict future depression status. Thus, the goal of this specific application is to test a comprehensive model of age-related changes to brain circuitry, neurocognitive performance, and social support as predictors of emotion regulation abilities and depressive symptoms in individuals with and without MDD. Reappraisal and distraction are the emotion regulation strategies of primary interest.

Models will be evaluated using primarily a series of linear (multiple) regression models focusing on between-subject effects/comparisons (age, MDD status, etc.) and the emotion regulation outcomes separately for reappraisal and distraction processes. As an extension of these models we will perform Structural Equation Modeling (SEM) type modeling to summarize the liability dimensions underlying the specific domains of depression [BDI scores measuring depression severity; lifetime duration of depressive episode(s)], and neural measures of dorsal attention network functioning [gPPI connectivity between dlPFC and amygdala; task-based activation during distraction in dACC, dlPFC, and inferior parietal lobe; DTI FA measure in SLF II] and affective network functioning [gPPI connectivity between vlPFC and amygdala; task-based activation during reappraisal in vmPFC, vlPFC, and amygdala; DTI FA measure of UF]. The SEM will be especially useful in predicting the future depression that will be assessed at one-year follow up, where the predicted (best linear unbiased predictors-BLUPS) values of lower-dimensional latent traits, along with emotion regulation outcomes, can be used as predictors for future depression. Moreover, hierarchical modeling structures can be imposed on latent traits conditionally on a shared latent trait describing associations among several latent traits thus further reducing underlying dimensionality and simplifying computations. This single trait can be thought as a cumulative effect of all latent traits and can be used a single index of uncertainty in predicting future depression symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* age 35-75
* No MRI contra-indications (e.g., metal in body)
* Not currently pregnant
* Ambulatory
* No known uncorrected sensory deficits
* Estimated verbal IQ of 85+ as indicated by the North American Adult Reading test MDD group: Current MDD assessed by history of MDD as assessed by standardized SCID interview
* Control Group: no lifetime of history of MDD as assessed by standardized SCID interview

Exclusion Criteria:

* History of moderate or severe substance dependence, as assessed by standardized SCID interview
* History of psychosis, mania, or eating disorders, as assessed by standardized SCID interview
* Disorders with impact on brain characteristics (e.g., epilepsy, Parkinson's Disease) or history of stroke
* Contraindications to MRI scanning, as indicated on the MRI safety screening questionnaire
* Use of antidepressants or other psychotropics other than sleep aids in the past 4 weeks (8 weeks for fluoxetine)
* Indication of mild cognitive impairment or dementia. To meet screening criteria, participants must meet all of the following:

  * Scoring of 24 or higher on the Montreal Cognitive Assessment;
  * perform above 1.5 standard deviations on the following measures: HVLT delayed recall, Trail Making B, and Animal Naming based normative values

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 MDD and 100 non-depressed (ND) adult qualifying participants ranging in age from 35-75
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Success of emotion regulation strategy use. | baseline
  Self-reported negative affect and arousal following the use of reappraisal and distraction strategies
Depression symptom severity | 6 months
  Severity of depressive symptoms as measured by self report
Depression symptom severity | 12 months
  Severity of depressive symptoms as measured by self report

CONTACTS AND LOCATIONS:
Overall Officials: Moria Smoski, PhD, Principal Investigator — Duke Department of Psychiatry
Locations (2):
- United States (2):
  - Civitan Building, Duke Psychiatry and Behavioral Sciences, Durham, North Carolina
  - Psychiatry and Behavioral Services, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
This study qualifies as a NDA data sharing study under NIMH guidelines, therefore data will be shared to NDCT.

REFERENCES:
- [Background] Nienhuis FJ, van de Willige G, Rijnders CA, de Jonge P, Wiersma D. Validity of a short clinical interview for psychiatric diagnosis: the mini-SCAN. Br J Psychiatry. 2010 Jan;196(1):64-8. doi: 10.1192/bjp.bp.109.066563. PMID 20044664
- [Background] Winecoff A, Labar KS, Madden DJ, Cabeza R, Huettel SA. Cognitive and neural contributors to emotion regulation in aging. Soc Cogn Affect Neurosci. 2011 Apr;6(2):165-76. doi: 10.1093/scan/nsq030. Epub 2010 Apr 12. PMID 20385663
- [Background] Levenson RW, Carstensen LL, Friesen WV, Ekman P. Emotion, physiology, and expression in old age. Psychol Aging. 1991 Mar;6(1):28-35. doi: 10.1037//0882-7974.6.1.28. PMID 2029364
- [Background] Knight BG, Maines ML, Robinson GS. The effects of sad mood on memory in older adults: a test of the mood congruence effect. Psychol Aging. 2002 Dec;17(4):653-61. doi: 10.1037//0882-7974.17.4.653. PMID 12507361